CLINICAL TRIAL: NCT00359489
Title: A Randomized, Open-Label, Methodology Trial To Investigate The Utility Of Echocardiography In Assessment Of Cardiac Valvular Regurgitation In Adult Subjects
Brief Title: Methods Study to Evaluate Use of Cardiac Ultrasound to Assess Heart Valve Abnormality in People.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Other Study IDs: A9001336
Record Dates: First submitted 2006-07-31; First posted 2006-08-02 (Estimated); Last update posted 2007-09-17 (Estimated); Status verified 2007-09

CONDITIONS: Heart Valve Diseases
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Device: cardiac echosonography

SUMMARY:
Methods study to evaluate use of cardiac ultrasound to assess heart valve abnormality in people.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years of age subjects with stable concomitant diseases with BMI >=30 kg/m2

Exclusion Criteria:

* Pregnant females
* Those with unstable/new onset diseases
* Those who are on agents known to be associated with cardiac valvular heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2007-04; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9001336&StudyName=Methods%20study%20to%20evaluate%20use%20of%20cardiac%20ultrasound%20to%20assess%20heart%20valve%20abnormality%20in%20people.%20%20